CLINICAL TRIAL: NCT03527212
Title: A Double-Masked, Randomized, Multicenter, Placebo-Controlled, Parallel-Group Study to Assess the Safety and Efficacy of SJP-0035 0.001% for the Treatment of Patients With Dry Eye Disease (DELTA-1 Study)
Brief Title: A Study to Assess the Safety and Effectiveness of SJP-0035 for the Treatment of Patients With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Senju Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJP-0035/3-01
Record Dates: First submitted 2018-05-04; First posted 2018-05-17 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Dry Eye Syndromes
Keywords: Dry Eye Disease; Corneal Epithelial Disorders; Re-Epithelialization
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SJP-0035 0.001% (ophthalmic solution) (Experimental)
  Interventions: Drug: SJP-0035 0.001%
- Placebo (ophthalmic solution) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SJP-0035 0.001% — Self-administration of 1 drop (approximately 40 µL) of 0.001% SJP-0035 ophthalmic solution into each eye 4 times daily for 4 weeks
  Arms: SJP-0035 0.001% (ophthalmic solution)
Drug: Placebo — Self-administration of 1 drop (approximately 40 µL) of placebo ophthalmic solution into each eye 4 times daily for 4 weeks
  Arms: Placebo (ophthalmic solution)

SUMMARY:
A double-masked, randomized, multi-center, placebo-controlled, parallel-group study in adult patients with Dry Eye Disease (DED). Patients will be randomly assigned to receive either SJP-0035 0.001% or placebo

DETAILED DESCRIPTION:
There are currently no approved products available anywhere worldwide for the treatment of Dry Eye Disease (DED) that directly affect the corneal epithelium. This study will evaluate the safety and efficacy of SJP-0035 0.001%, compared with a placebo, on corneal healing. Patients meeting the requirements of the inclusion/exclusion criteria will administer 1 drop of the study drug/placebo 4 times per day for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF).
* Has Dry Eye Disease (DED) with moderate to severe corneal fluorescein staining in both eyes.
* Has blurred vision caused by DED in both eyes.
* Women of childbearing potential must have negative serum pregnancy test results at Screening and Randomization and agree to use effective contraception throughout the study; post-menopausal women must have negative serum pregnancy test results at Screening and Randomization.
* Male participants must agree to use an acceptable form of contraception (i.e. a condom plus spermicide) and to refrain from sperm donation throughout the study.

Exclusion Criteria:

* Has any corneal stromal or endothelial abnormalities in either eye.
* Has any active or chronic allergic, bacterial or viral infection of ocular adnexa and eye structures in either eye.
* Has had eye surgery (including cataract, vitreous or eyelid surgery) in either eye within the last 28 days prior to first dose of study drug.
* Has had refractive surgery (including eye surface laser surgery) in either eye within the last 180 days prior to first dose of study drug.
* Has used any eye medication in either eye within 14 days prior to first dose of study drug, or is anticipated to require such medications during the study. Preservative-free artificial tears may be used up to 72 hours prior to the first dose in either eye.
* Is a contact lens wearer and cannot discontinue use in both eyes from Screening through the duration of the study.
* Has previously received SJP-0035 (study drug) in either eye.
* Currently has punctal occlusions, of any type, inserted into both superior and inferior puncta in either eye at Screening through the duration of the study.

Other protocol-defined inclusion/exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Corneal fluorescein staining | Week 5
  Number of patients showing complete clearing of corneal fluorescein staining, scored on the Baylor grading system.

SECONDARY OUTCOMES:
Blurred vision | Week 5
  Improvement in blurred vision from baseline, using a 100-point visual analog score (VAS) where 0 indicates no blurred vision and 100 indicates the worst possible blurred vision.

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Arizona Eye Center, 1500 West Ray Road, Chandler, Arizona
  - Walman Eye Center, 10615 West Thunderbird Boulevard, Suite D180, Sun City, Arizona
  - SoCal Eye Physicians and Associates Surgery Center, 3300 E. South Street, Long Beach, California
  - East West Eye Institute, 420 East 3rd Street, Suite 603, Los Angeles, California
  - North Valley Eye Medical Group, Inc., Suite 341, 11550 Indian Hills Road, Mission Hills, California
  - North Bay Eye Associates, Inc., 104 Lynch Creek Way, Petaluma, California
  - Sibia Eye Institute, Suite 1 & 2, 11195 Jog Road, Boynton Beach, Florida
  - Clayton Eye Center, Suite 100 and 120, 1000 Corporate Center Drive, Morrow, Georgia
  - Coastal Research Associates, LLC., Suite J3, 11205 Alpharetta Highway, Roswell, Georgia
  - Chicago Cornea Consultants, Ltd., Suite 502, 1585 North Barrington Road, Hoffman Estates, Illinois
  - The Eye Care Institute, 1536 Story Avenue, Louisville, Kentucky
  - Chu Vision Institute, 9117 Lyndale Avenue South, Bloomington, Minnesota
  - Tauber Eye Center, Suite 202, 4400 Broadway, Kansas City, Missouri
  - Emil A. Stein, M.D., Ltd., Suite 100, 2090 East Flamingo Road, Las Vegas, Nevada
  - Ophthalmic Consultants of Long Island, 3rd Floor, 360 Merrick Road, Lynbrook, New York
  - South Shore Eye Care LLC, 2185 West Wantagh Avenue, Wantagh, New York
  - Cornerstone Eye Care, High Point, North Carolina
  - Black Hills Regional Eye Institute, 2800 3rd Street, Rapid City, South Dakota
  - Hill Country Eye Center, Cedar Park, Texas
  - Alkek Eye Center, 1977 Butler Boulevard, Houston, Texas
  - R and R Eye Research, LLC., Suite 100, 5430 Fredericksburg Road, San Antonio, Texas
  - Southern Utah Medical Research, Suite 100, 292 South 1470 East, St. George, Utah
  - Virginia Eye Consultants, 241 Corporate Boulevard, Norfolk, Virginia

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls